CLINICAL TRIAL: NCT00214747
Title: An Imaging Trial of the Distribution of Topical Gel Formulations in the Human Vagina: Candidate Formulations
Brief Title: An Imaging Trial of the Distribution of Topical Gel Formulations in the Human Vagina
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biosyn (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: RRU-003
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-10-25 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: Vehicle gel formulations

SUMMARY:
This study is designed to assess the distribution and spread of four different vehicle formulations in the vagina. In-vivo data will be obtained regarding each vehicle formulation at various time points after insertion of the gel into the vagina.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 year old women
* non-pregnant
* healthy

Exclusion Criteria:

* abnormal finding on pelvic exam
* pregnant or breastfeeding
* allergy to intravaginal products
* history of claustrophobia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6
Dates: Start 2005-03; Study Completion 2005-11

PRIMARY OUTCOMES:
MRI evaluation of gel formulation distribution in vagina
Total linear distance in mm covered by gel
Surface area actually covered by gel (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Barnhart, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Rreproductive Research Unit, U of Penn Medical Center, Philadelphia, Pennsylvania, United States